CLINICAL TRIAL: NCT02000999
Title: The Diagnostic Yield of Malignancy Comparing Cytology, FISH and Molecular Analysis of Cell Free Cytology Brush Supernatant in Patients With Biliary Strictures Undergoing Endoscopic Retrograde Cholangiography (ERC): A Prospective Study
Brief Title: Diagnosis of Bile Duct Strictures
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Cytology 2013-201211068
Record Dates: First submitted 2013-11-19; First posted 2013-12-04 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Bile Duct Stricture; Cholangiocarcinoma; Pancreatic Cancer; Chronic Pancreatitis
Keywords: Bile duct stricture; Cholangiocarcinoma; Pancreatic cancer; Chronic pancreatitis
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Pancreatitis, Chronic | interventions — Cytological Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with bile duct strictures
  Interventions: Other: brushing of bile duct strictures for cytology

INTERVENTIONS:
Other: brushing of bile duct strictures for cytology

SUMMARY:
The purpose of this prospective study is to compare the diagnostic utility of two techniques (brush cytology + FISH and brush cytology + free DNA analysis) in the diagnosis of biliary strictures. Histologic diagnosis (biopsies) in conjunction with clinical and/or imaging follow-up will serve as the gold standard for diagnosis of malignancy. In order to do this the investigators will ask study participants to have a small volume of fluid obtained from the bile duct sent for additional testing at RedPATH. In some patients additional brushings will be obtained for FISH testing (this adds <2 minutes to ERCP and only associated risk is increased procedure duration).

The investigators hypothesize that the use of cytology +DNA analysis has a higher sensitivity and accuracy when compared to cytology +FISH in patients with biliary strictures.

Primary aim:

To compare the sensitivity and accuracy of the two techniques (brush cytology + FISH and brush cytology + free DNA analysis). Histologic diagnosis (histology from biopsy or cytology for fine needle aspiration) in conjunction with clinical and/or imaging follow-up will serve as the gold standard for diagnosis of malignancy.

Secondary aims:

1. To evaluate the diagnostic yield of malignancy when all three techniques (cytology, FISH and DNA analysis) are used.
2. To evaluate the added value of biliary forceps biopsies, when used in conjunction with cytology, FISH and DNA analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age: > 18 years
2. Presence of a biliary stricture
3. Ability to provide written informed consent.

Exclusion Criteria:

1. Severe coagulopathy (INR > 1.8) or thrombocytopenia (platelet count <50,000)
2. Inability to cannulate the common bile duct
3. Presence of altered anatomy (Billroth II or Roux-en-Y reconstruction)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 undergoing ERCP for the diagnosis and treatment of bile duct stricture
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2013-11; Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
• Sensitivity accuracy of cytology, FISH and mutation profiling using histologic diagnosis in conjunction with clinical and/or imaging follow-up as the gold standard. | 2 years

SECONDARY OUTCOMES:
• Specimen adequacy | 2 years
• Complications (pancreatitis, bleeding, perforation, cholangitis) | 2 years
• Technical success and ease of procedure | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States